CLINICAL TRIAL: NCT06664086
Title: Economic and Psychological Burden of Infertility Among Women Attending Women Health Hospital, Assiut University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abdelmalek Abdallah, assistant lecturer, Assiut University
Other Study IDs: burden of infertility on women
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Burden, Infertility
MeSH Terms: conditions — Infertility | interventions — Economics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infertile women: women suffering from infertility
  Interventions: Behavioral: economic and psychological burden
- fertile women: women having children not suffering from infertility.
  Interventions: Behavioral: economic and psychological burden

INTERVENTIONS:
Behavioral: economic and psychological burden — measuring the economic and psychological burden of infertility

SUMMARY:
Rational of the study:

Infertility is a significant reproductive health issue for couples worldwide. The effects of infertility are wide-ranging-from mental health issues such as anxiety and depression to social and economic issues such as ostracization and economic problems. Although infertility affects both men and women, the woman in a couple is most often blamed for the inability to bear children.

DETAILED DESCRIPTION:
Infertility is a disease of the male or female reproductive system, defined by the failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourse (WHO).

Large numbers of people are affected by infertility in their lifetime, according to a new report published by World Health Organization. Around 17.5% of the adult population - roughly 1 in 6 worldwide - experience infertility. The inability to conceive children is experienced as a stressful situation by individuals and couples all around the world. The consequences of infertility are manifold and may include societal repercussions and personal emotional suffering. The infertile couple experienced greater dissatisfaction with themselves and their marriages. Females experienced greater discontent over time and had greater emotional problems than males because infertility had traditionally been viewed as a women problem and women have been expected to suffer greater emotional problems due to infertility. Treatment for infertility provides an opportunity for women and men to become parents. The evolution of assisted reproductive technology (ART) for the treatment of infertile couples is considered an extraordinary restorative accomplishment throughout the world. However accessibility of treatments such as IVF is limited to only those who can afford to pay out of pocket (OOP). Even among those who have the ability to pay, their willingness and financial ability to undergo multiple cycles of ART often depends on OOP payments incurred. However, due to the desire for a child, couples are often ready to make significant financial sacrifices often beyond their means. Couples are frequently willing to suffer catastrophic financial hardship instead of forgoing infertility care, resulting in negative economic consequences. Evidence suggests that in the absence of mechanisms for risk protection, OOP payments can push households into poverty.

ELIGIBILITY:
Inclusion Criteria:

* • reproductive age group 15 - 49

  * Duration of marriage not less than 1 year.
  * Has regular sexual intercourse without the functional use of contraceptive methods.
  * Free from any other debilitating chronic illness.

Exclusion Criteria:

* Women who have any previous psychological disease or treatment

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Data will be collected through a semi-structured interviewer administered questionnaire. From IVF unit and outpatient gynecological clinic at women health hospital, Assiut university .
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychological disorders as: anxiety, depression and stress among infertile women. | baseline
  measuring prevalence of psychological disorders as: anxiety, depression and stress among infertile women using DASS scale
Financial and economic suffering of infertile couples | baseline
  Financial and economic suffering of infertile couples

CONTACTS AND LOCATIONS:
Overall Officials: Omaima ELGibaly, Professor, Study Director — Professor at Public Health and Community Medicine Faculty of Medicine- Assiut University

REFERENCES:
- [Background] Poddar S, Sanyal N, Mukherjee U. Psychological profile of women with infertility: A comparative study. Ind Psychiatry J. 2014 Jul-Dec;23(2):117-26. doi: 10.4103/0972-6748.151682. PMID 25788801
- [Background] Dyer SJ, Sherwood K, McIntyre D, Ataguba JE. Catastrophic payment for assisted reproduction techniques with conventional ovarian stimulation in the public health sector of South Africa: frequency and coping strategies. Hum Reprod. 2013 Oct;28(10):2755-64. doi: 10.1093/humrep/det290. Epub 2013 Jul 21. PMID 23878180